CLINICAL TRIAL: NCT06640712
Title: The Evaluation of Oral and Dental Health in Substance Dependent Individuals
Brief Title: Oral and Dental Health in Substance Dependent Individuals
Acronym: ODH_SUD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Democracy University (Other)
Responsible Party: Principal Investigator, Hasan Tahsin Kilic, Asistant Profesor, Buca Seyfi Demirsoy State Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024/234
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Substance Use Disorder (SUD); Decayed Teeth; Teeth Loss; Teeth Missing
Keywords: substance use disorder; Oral health; DMTF index; Oral health behaviors
MeSH Terms: conditions — Substance-Related Disorders; Dental Caries; Anodontia | interventions — Metabolism

STUDY DESIGN:
Intervention Model Description: his study uses a parallel design to compare the oral health status among individuals with different substance use disorders (Methamphetamine, Cannabis, Polysubstance) and a healthy control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm 1: Methamphetamine Use Group (Experimental): This group consists of individuals diagnosed with Methamphetamine Use Disorder. Diagnoses were conducted by the same psychiatrist for all participants. Following psychiatric evaluation, participants underwent a clinical oral health examination to assess their dental health status, with the Decayed, Missing, and Filled Teeth (DMFT) index being calculated afterward. This group is included to investigate the impact of methamphetamine use on oral health.
  Interventions: Diagnostic Test: Dental caries was assessed using the DMFT index (Decayed, Missing, and Filled Teeth) according to the World Health Organization's caries diagnostic criteria.; Diagnostic Test: Substance Use Disorder Diagnosis
- Arm 2: Cannabis Use Group (Experimental): This group consists of individuals diagnosed with Cannabis Use Disorder. Diagnoses were performed by the same psychiatrist for consistency. After the psychiatric assessment, participants received a clinical oral health examination to determine their dental health status, and the DMFT index was calculated subsequently. This group aims to assess the effects of cannabis use on oral health.
  Interventions: Diagnostic Test: Dental caries was assessed using the DMFT index (Decayed, Missing, and Filled Teeth) according to the World Health Organization's caries diagnostic criteria.; Diagnostic Test: Substance Use Disorder Diagnosis
- Arm 3: Polysubstance Use Group (Experimental): This group includes individuals who use multiple substances (polysubstance use disorder). All participants were evaluated by the same psychiatrist to ensure diagnostic accuracy. Following their psychiatric evaluation, participants had a clinical oral health examination, during which the DMFT index was calculated to assess dental health. This group is included to examine the impact of polysubstance use on oral health.
  Interventions: Diagnostic Test: Dental caries was assessed using the DMFT index (Decayed, Missing, and Filled Teeth) according to the World Health Organization's caries diagnostic criteria.; Diagnostic Test: Substance Use Disorder Diagnosis
- Arm 4: Control Group (Other): Healthy, non-substance-using individuals This group consists of healthy individuals with no history of substance use, systemic medical conditions, or regular medication use. Diagnoses were confirmed by the same psychiatrist. Afterward, participants underwent a clinical oral health examination, and the DMFT index was calculated to provide a baseline for comparison with substance-using groups. This group serves as the control group to compare the dental health outcomes of non-substance-using individuals.
  Interventions: Diagnostic Test: Dental caries was assessed using the DMFT index (Decayed, Missing, and Filled Teeth) according to the World Health Organization's caries diagnostic criteria.

INTERVENTIONS:
Diagnostic Test: Dental caries was assessed using the DMFT index (Decayed, Missing, and Filled Teeth) according to the World Health Organization's caries diagnostic criteria. — The same psychiatrist administered the Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) to all participants. Oral health examinations were performed by a trained dental student and a specialist dentist using a portable dental chair, artificial light, and a dental mirror. Dental caries was assessed using the DMFT index (Decayed, Missing, and Filled Teeth) according to the World Health Organization's caries diagnostic criteria. This index included the number of decayed, missing (due to caries, excluding 3rd molars), and filled teeth in the permanent dentition. The oral health examiners were blinded to each participant's substance use type and sociodemographic information.
Diagnostic Test: Substance Use Disorder Diagnosis — This intervention involves a psychiatric evaluation conducted by a licensed psychiatrist to diagnose Substance Use Disorder according to the criteria outlined in the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5). The psychiatrist performs a comprehensive assessment of each participant's substance use history and related behaviors. This diagnosis step is essential for identifying participants with specific substance use disorders, such as Methamphetamine, Cannabis, or Polysubstance Use Disorders, before proceeding with the dental health examination.
  Arms: Arm 1: Methamphetamine Use Group; Arm 2: Cannabis Use Group; Arm 3: Polysubstance Use Group

SUMMARY:
The goal of this cross-sectional clinical study is to compare the oral health status of individuals with Methamphetamine (MA), Cannabis (THC), and Polysubstance (PSU) use disorders to healthy controls. The study aims to answer:

How does substance use type (Methamphetamine, Cannabis, Polysubstance) affect dental health outcomes as measured by the DMFT index? What is the relationship between substance use characteristics (type, duration, and quantity) and oral health behaviors? Researchers will compare individuals with substance use disorders to a control group of healthy, non-substance-using individuals to assess the impact of different substances on dental health.

Participants will:

Undergo a clinical oral examination to evaluate dental health using the DMFT index.

Complete a questionnaire on sociodemographic information, substance use history, and oral health behaviors based on the Hiroshima University Dental Behavior Inventory (HU-DBI).

This study contributes to understanding the dental health needs of individuals with substance use disorders and the importance of tailored dental interventions for this population.

DETAILED DESCRIPTION:
This cross-sectional clinical study was conducted at İzmir Democracy University Buca Seyfi Demirsoy Education and Research Hospital Probation Clinic from April to August 2024. In line with Turkish policy, individuals involved in substance-related offenses attended probation clinics, where this study's participants were recruited. A sample of 190 individuals with Methamphetamine (MA), Cannabis (THC), and Polysubstance (PSU) use disorders was compared to a control group of 91 healthy male hospital employees with no history of substance use.

All participants underwent clinical oral health examinations performed by a trained dental student and specialist dentist, assessing dental health using the Decayed, Missing, and Filled Teeth (DMFT) index based on WHO diagnostic criteria. The clinical assessments were conducted with a portable dental chair, artificial lighting, and a dental mirror. The examiners were blinded to participants' substance use and sociodemographic details.

In addition to clinical examinations, sociodemographic data, substance use history, and oral health behaviors were collected through a researcher-developed questionnaire and the Turkish version of the Hiroshima University Dental Behavior Inventory (HU-DBI). The study aimed to identify differences in dental health outcomes across substance use groups and to assess the relationships between oral health and variables such as substance type, usage duration, and oral health behaviors.

Statistical analyses were conducted using SPSS 26.0, applying t-tests, ANOVA, Chi-square tests, and Pearson correlation to evaluate differences and correlations across variables. A significance level of p<0.05 was applied for all tests. The findings contribute to understanding the dental health needs of individuals with substance use disorders, underscoring the importance of targeted dental care interventions for this population.

ELIGIBILITY:
Inclusion Criteria:

* Male participants
* aged 18 to 45
* methamphetamine, cannabis, or polysubstance users.

Exclusion Criteria:

* absence of urine toxicology analysis results,
* use of substances other than methamphetamine or cannabis,
* being under the influence of substances during the evaluation
* not meeting DSM-5 criteria for Substance Use Disorder,
* having any systemic medical conditions
* current medication use
* incomplete scales and forms.
* who wore removable dentures
* In the control group, individuals with a history of any substance use

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 281 (Actual)
Dates: Start 2024-04-25 (Actual); Primary Completion 2024-08-25 (Actual); Study Completion 2024-08-25 (Actual)

PRIMARY OUTCOMES:
Compare the oral health status of individuals with Methamphetamine (MA), Cannabis (THC), and Polysubstance (PSU) Use Disorders to healthy controls assessed by DMFT index | Up to 24 weeks
  Dental caries was assessed using the DMFT index (Decayed, Missing, and Filled Teeth) according to the World Health Organization's caries diagnostic criteria. This index included the number of decayed, missing (due to caries, excluding 3rd molars), and filled teeth in the permanent dentition. A minimum score of 0 and a maximum score of 28 can be obtained on the DMFT scale, with higher scores indicating poorer oral health.

CONTACTS AND LOCATIONS:
Overall Officials: Osman HT Kılıç, Asist. Prof., Study Director — Izmir Democracy University
Locations (1):
- İzmir Demokrasi Üniversitesi, Izmir, Konak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Due to the sensitive nature of the data, individual participant data (IPD) will be shared only with researchers who sign a data use agreement. This agreement will stipulate the purpose of data usage, ensuring that the data will be used solely for scientific research and not for any non-research purposes.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The IPD and supporting information will be available after the study has been published in an international peer-reviewed journal and will remain accessible for five years following publication.
Access Criteria: ccess will be granted to qualified researchers who provide a scientific rationale for data usage and agree to sign a data use agreement. This agreement will stipulate that the data will be used exclusively for scientific research purposes

REFERENCES:
- [Derived] Kilic OHT, Kurklu Arpacay D, Gezen OC, Bayram ZN, Baser A. Comparative effects of methamphetamine, cannabis, and polysubstance use on oral health. Front Psychiatry. 2025 Jan 31;16:1510228. doi: 10.3389/fpsyt.2025.1510228. eCollection 2025. PMID 39958156
- See also: The study was conducted at the İzmir Democracy University Buca Seyfi Demirsoy Education and Research Hospital's Probation Clinic (Denetimli Serbestlik Polikliniği). This clinic provides treatment and evaluation services for individuals who have been man — https://bucadh.saglik.gov.tr/TR-998180/denetimli-serbestlik-poliklinigi.html